CLINICAL TRIAL: NCT02686372
Title: A Phase I Study of T Cell Receptor-Redirected T Cell Infusion For Prevention of Hepatocellular Carcinoma Recurrence in Subjects With Hepatitis B Virus-Related Hepatocellular Carcinoma Post Liver Transplantation
Brief Title: A Study of TCR-Redirected T Cell Infusion to Prevent Hepatocellular Carcinoma Recurrence Post Liver Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lion TCR Pte. Ltd. (Industry)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: LTCR-HCC-1-1
Record Dates: First submitted 2016-02-17; First posted 2016-02-19 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; hepatitis B virus-related; post liver transplantation; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBV/TCR-T cell infusion (Experimental): Subjects enrolled in the experimental (treatment) group will receive escalating doses of HBV/ TCR expressing autologous T cells. The interval between the first two doses is 14 days, followed by one month of safety monitoring, before subsequent two doses of 1 month interval in between. Thereafter, subjects would enter into observation period of the safety and tolerability of the treatment and will be followed up until disease relapse.
  Interventions: Biological: TCR-T
- No intervention and TCR-T (at crossover) (Other): No intervention and to be crossover to experimental arm upon confirmation of disease recurrence.
  Interventions: Biological: No intervention and TCR-T (at crossover)

INTERVENTIONS:
Biological: TCR-T — Autologous T cells transfected with mRNA encoding HBV antigen-specific TCR
  Arms: HBV/TCR-T cell infusion
Biological: No intervention and TCR-T (at crossover) — Autologous T cells transfected with mRNA encoding HBV antigen-specific TCR
  Arms: No intervention and TCR-T (at crossover)

SUMMARY:
Hepatocellular Carcinoma (HCC) recurrence rate is high among liver transplant patients, while treatment measures are limited. This study plans to recruit 39 subjects with Hepatitis B virus (HBV) related HCC after liver transplantation. The objective of the study is to assess the safety, tolerability and effectiveness of the HBV specific T cell receptor (HBV/TCR) redirected T cell in the target population.

DETAILED DESCRIPTION:
A open-label, cohort clinical study of T cell receptor-redirected T cells to prevent recurrence of HBV-related hepatocellular carcinoma after liver transplantation. Subjects will be enrolled into the observation cohort or treatment cohort.

Subjects enrolled in the treatment group will receive escalating doses of HBV/ TCR expressing autologous T cells after confirming eligibility. The interval between the first two doses is 14 days, followed by one month of safety monitoring, before subsequent two doses of 1 month interval in between. Thereafter, subjects would enter into observation period of the safety and tolerability of the treatment and will be followed up until disease relapse.

Upon disease recurrence, eligible patient may receive HBV specific T-cell receptor (TCR-T) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as hepatocellular carcinoma (HCC)
* Underwent liver transplantation
* Seropositive for hepatitis B surface antigen (HBsAg), or presence of HBV DNA or HBV RNA before liver transplantation
* Expression of TCR-T target epitopes within specific human leukocyte antigen (HLA) class I profile
* No major post-operative complication
* Life expectancy of at least 3 months
* Ability to provide informed consent
* Ability to comply with study procedures

Exclusion Criteria:

* Known, clinically suspected or has history or central nervous system (CNS) and bone metastasis
* Significant ongoing immunologic rejection based on pathology and clinical diagnosis
* Evidence or history of significant bleeding diathesis or coagulopathy
* Prior exposure to any cell therapy such as, but not limited to NK, CIK, DC, CTL, stem cells therapy
* Known history of testing positive for human immunodeficiency virus (HIV) 1 or 2 or known acquired immunodeficiency syndrome (AIDS)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Women who are pregnant or breast-feeding
* Any condition that is unstable or which could jeopardise the safety of the patient and his/her compliance in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
To Evaluate safety of the TCR-T treatment | Start of Treatment until 28 days post last dose
  Measures include
  - assessments of Adverse Events (AEs) and Serious AEs,

SECONDARY OUTCOMES:
To evaluate Progression Free Survival rate | Start of Treatment until disease progression, and subsequent follow up for 2 years or death (whichever comes first)
  PFS
To evaluate Duration of response rate | Start of Treatment until disease progression, and subsequent follow up for 2 years or death (whichever comes first)
  DOR
To evaluate objective response rate | Start of Treatment until disease progression, and subsequent follow up for 2 years or death (whichever comes first)
  ORR

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoshun He, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun-Yat Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qasim W, Brunetto M, Gehring AJ, Xue SA, Schurich A, Khakpoor A, Zhan H, Ciccorossi P, Gilmour K, Cavallone D, Moriconi F, Farzhenah F, Mazzoni A, Chan L, Morris E, Thrasher A, Maini MK, Bonino F, Stauss H, Bertoletti A. Immunotherapy of HCC metastases with autologous T cell receptor redirected T cells, targeting HBsAg in a liver transplant patient. J Hepatol. 2015 Feb;62(2):486-91. doi: 10.1016/j.jhep.2014.10.001. Epub 2014 Oct 13. PMID 25308176
- [Background] Gehring AJ, Xue SA, Ho ZZ, Teoh D, Ruedl C, Chia A, Koh S, Lim SG, Maini MK, Stauss H, Bertoletti A. Engineering virus-specific T cells that target HBV infected hepatocytes and hepatocellular carcinoma cell lines. J Hepatol. 2011 Jul;55(1):103-10. doi: 10.1016/j.jhep.2010.10.025. Epub 2010 Nov 23. PMID 21145860
- [Background] Koh S, Shimasaki N, Suwanarusk R, Ho ZZ, Chia A, Banu N, Howland SW, Ong AS, Gehring AJ, Stauss H, Renia L, Sallberg M, Campana D, Bertoletti A. A practical approach to immunotherapy of hepatocellular carcinoma using T cells redirected against hepatitis B virus. Mol Ther Nucleic Acids. 2013 Aug 13;2(8):e114. doi: 10.1038/mtna.2013.43. PMID 23941866